CLINICAL TRIAL: NCT07392749
Title: Feasibility Study of Diaphragm Synchronized Pacing (DSP) Via the Left Inferior Phrenic Vein (LIPV) Approach
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Tianbao Yao, Associate Chief Physician, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSP-LIPV study
Record Dates: First submitted 2025-12-08; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: CRT; CRT-D; DSP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DSP LIPV group (Experimental)
  Interventions: Procedure: DSP

INTERVENTIONS:
Procedure: DSP — For patients with indications for CRT or CRT-D, a pacing electrode delivery sheath is inserted via the subclavian approach following the placement of the atrial electrode as part of the conventional pacemaker implantation procedure. Angiography is performed at the level of the LIPV to visualize its course. Subsequently, a quadripolar ventricular lead is advanced through the sheath into the LIPV to conduct diaphragmatic pacing testing, observing the diaphragmatic pacing effectiveness and its impact on cardiac activity. Upon test completion, the catheter and lead are withdrawn, and the standard pacemaker implantation procedure is continued.

SUMMARY:
Cardiac resynchronization therapy（CRT） benefits a portion of patients, while more patients are not yet indicated to a therapy that mechanically helps the heart systole and/or diastole. Synchronized diaphragmatic pacing may be feasible to induce diaphragm local contraction and recoil that enhance pump function of the heart, thus improve cardiac function and QoL.

This acute, interventional study is conducted in a single site, Renji Hospital, to evaluate the feasibility of diaphragm pacing and assess the beneficial effect of pacing-regulated diaphragm movement to the heart, with 10 cases of sample size and one-week follow-up after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >=18 yrs;
* Patients indicated for CRT or CRT-D , planned for LV lead implantation;
* Patients are willing to participate in the study and provide signed informed consent

Exclusion Criteria:

* CRT or CRT-D replacement
* Ischemic heart disease with CABG history
* Diaphragm dysfunction history
* Phrenic nerve injury
* IVC filter history
* Abdominal surgery history
* Splenomegaly
* Pulmonary disease
* Moderate or severe liver cirrhosis
* Severe hepatic or renal dysfunction
* Currently pregnant or planning pregnancy during the study period
* Patients participate in another study that will confound this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The feasibility of local diaphragm muscle pacing | Acute, during the procedure
  To evaluate the success rate of diaphragm pacing and the capability of the electrode to capture the local diaphragm below the cardiac apex, providing a recommendation of venous access and route for the interventional procedure to conduct local electrical stimulation in the diaphragm.

SECONDARY OUTCOMES:
The observation of pacing-regulated diaphragm movement for the determination of local diaphragm capture | Intra-procedure
The diameter (or dimension) of the local venous anatomy | Perioperative
DSP lead threshold | Intra-procedure
Complications of the diaphragmatic synchronized pacing | Perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Dando L, Howick V JF, Yoo J, Kella DK, McLeod CJ, van Niekerk CJ. Left inferior phrenic vein ICD lead implantation. HeartRhythm Case Rep. 2025 Mar 18;11(6):534-538. doi: 10.1016/j.hrcr.2025.03.010. eCollection 2025 Jun. No abstract available. PMID 40557395
- [Background] McIntosh RA, Ansari MI, Moon J, Khan HR. Delivery of cardiac resynchronization therapy via the left inferior phrenic vein: a case report. Eur Heart J Case Rep. 2019 Sep 16;3(3):ytz144. doi: 10.1093/ehjcr/ytz144. eCollection 2019 Sep. PMID 31660505
- [Background] Fujii Y, Koizumi J, Sekiguchi Y, Ono S, Sekiguchi T, Hara T, Hashimoto J. Morphometric assessment of the left inferior phrenic vein in patients with portal hypertension. Sci Rep. 2022 Sep 10;12(1):15275. doi: 10.1038/s41598-022-19610-w. PMID 36088466
- [Background] Beeler R, Schoenenberger AW, Bauer P, Kobza R, Bergner M, Mueller X, Schlaepfer R, Zuber M, Erne S, Erne P. Improvement of cardiac function with device-based diaphragmatic stimulation in chronic heart failure patients: the randomized, open-label, crossover Epiphrenic II Pilot Trial. Eur J Heart Fail. 2014 Mar;16(3):342-9. doi: 10.1002/ejhf.20. Epub 2013 Dec 6. PMID 24464736
- [Background] Roos M, Kobza R, Jamshidi P, Bauer P, Resink T, Schlaepfer R, Stulz P, Zuber M, Erne P. Improved cardiac performance through pacing-induced diaphragmatic stimulation: a novel electrophysiological approach in heart failure management? Europace. 2009 Feb;11(2):191-9. doi: 10.1093/europace/eun377. PMID 19168496
- [Background] Sieniewicz BJ, Gould J, Porter B, Sidhu BS, Teall T, Webb J, Carr-White G, Rinaldi CA. Understanding non-response to cardiac resynchronisation therapy: common problems and potential solutions. Heart Fail Rev. 2019 Jan;24(1):41-54. doi: 10.1007/s10741-018-9734-8. PMID 30143910
- [Result] Jorbendaze A, Young R, Shaburishvili T, Demyanchuk V, Buriak R, Todurov B, Rudenko K, Zuber M, Stampfli SF, Tanner FC, Erne P, Mirro M, Fudim M, Goldberg LR, Cleland JGF. Synchronized diaphragmatic stimulation for heart failure using the VisONE system: a first-in-patient study. ESC Heart Fail. 2022 Aug;9(4):2207-2214. doi: 10.1002/ehf2.13984. Epub 2022 May 26. PMID 35619238